CLINICAL TRIAL: NCT06838312
Title: Reuse of Polyp Traps, a Way to Approach Sustainability: A Multicentric Non-inferiority Study
Brief Title: Reuse of Polyp Traps, a Way to Approach Sustainability
Acronym: POLYPTRAP
Status: Not yet recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Consorci Sanitari de Terrassa (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario La Fe (Other); Hospital Sant Bernabé de Berga (Unknown); Hospital Dos de Maig (Unknown); Hospital Universitari Joan XXIII de Tarragona. (Other); Centro Medico Teknon (Other); Clínica Mi Tres Torres Barcelona (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIBSP-RPT-2024-69
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cross Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reuse Group: patients from centres that routinely reuse polyp traps.
  Interventions: Other: Reuse or dispose a polyp trap
- Single Use Group: patients from centres that dispose polyp traps after a single use.
  Interventions: Other: Reuse or dispose a polyp trap

INTERVENTIONS:
Other: Reuse or dispose a polyp trap — Participant hospitals will be separated into two groups, according to their standard clinical practice: A) reuse or B) dispose polyp traps after a colonoscopy with polypectomy. Centres will participate with their current method of using polyp traps. Work dynamics will not change as patients will be recruited from centers that routinely reuse or dispose polyp traps.

SUMMARY:
The environmental impact of healthcare practice in the context of climate change is in the spotlight. Digestive endoscopy units are the third hospital unit that generates the most waste and environmental impact. For this reason, scientific societies advice studying and adopting more sustainable clinical practices, reconsidering current protocols for reprocessing and disinfection of single-use material. One of the devices, widely used and which generates a large amount of waste, is the polyp trap. It allows an easy recovery of the polyps removed during endoscopy. This device is discarded after a single use in some centers, and reused after washing and disinfection in others. Manufacturers recommend the single-use of the device, even there is no scientific evidence to support this action. In the investigators endoscopy unit, 3800 polyp traps are used yearly. The investigators hypothesis is that reusing the polyp catcher has similar safety to disposal after a single use, with better environmental and economic results. Objectives: To evaluate the safety of the reused and discarded after a single-use polyp trap. The investigators will assess 1) the post-colonoscopy infection rate and 2) the reliability of the anatomopathological study, 3) CO2 emissions and 4) costs of each practice. Methodology: A non-inferiority study will be carried out by observing the usual clinical practice of different centers and collecting data that suggest infection, cross-sampling and general complications. The results will be easily applicable in endoscopy units and will serve as a basis for future studies with other more controversial devices.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo an elective colonoscopy will be recruited for the study.

  * Written informed consent to participate in the study and willingness to be contacted by telephone for follow-up.

Exclusion Criteria:

* Patients who complete the colonoscopy without a polypectomy.
* Patients who complete the colonoscopy without the use of a polyp trap.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who have undergone a colonoscopy in which a polyp trap was used.
Sampling Method: Non-Probability Sample
Enrollment: 3238 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with symptoms suggesting infection | Follow up at day 15
  Did the patient present any of the following symptoms or diagnosis after the endoscopy?
  * Fever
  * Bacteraemia
  * Bronchoaspiration / Pneumonia
  * Other: Comments:
  * None
Number of infectious events related to endoscopy | Follow up at day 15
  Was the event related to the endoscopy procedure? Yes / Probably / Doubtfully / No
Number of infectious events related to polyp trap | Follow up at day 15
  Was the event related to the polyptrap? Yes / Probably / Doubtfully / No

SECONDARY OUTCOMES:
Number of inconsistent anatomopathological results | Follow up at day 15
  Was the anatomopathological finding consistent with the findings in the endoscopy?

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT06838312/Prot_SAP_000.pdf